CLINICAL TRIAL: NCT03551509
Title: Extracellular Matrix Scaffold Graft Augmentation in Rotator Cuff Repair: a Prospective, Randomized, Controlled Trial
Brief Title: LifeNet: Extracellular Matrix Graft in Rotator Cuff Repair
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor terminated early
Sponsor: Gregory Gilot (Other)
Collaborators: LifeNet Health (Industry); The Cleveland Clinic (Other)
Responsible Party: Sponsor-Investigator, Gregory Gilot, Staff Physician, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FLA 18-008
Record Dates: First submitted 2018-05-15; First posted 2018-06-11 (Actual); Results first posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Rotator Cuff Tear
Keywords: Rotator Cuff Tear; Large Rotator Cuff Tear; Massive Rotator Cuff Tear; ECM; Extracellular Matrix; ArthroFLEX
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Treatment Group (Active Comparator): Patients randomly assigned into the control group will undergo open or arthroscopic rotator cuff repair using the surgeon's standard practice. No ECM graft will be used.
  Interventions: Procedure: Control
- Treatment Group (Active Comparator): Patients randomly assigned into the treatment group will undergo open or arthroscopic rotator cuff repair with A-FLEX graft to augment the repair. ECM scaffold grafts are indicated for the reinforcement of soft tissues repaired by sutures or suture anchors during tendon repair surgery, including rotator cuff.
  Interventions: Procedure: ArthroFLEX ECM scaffold graft
- Alternative Treatment Group (Other): Patients who meet pre-op inclusion criteria where a repair cannot be accomplished due to intraoperative findings will remain in the study. This group will be analyzed separately and still follow study procedures.
  Interventions: Biological: Alternative Treatment Group

INTERVENTIONS:
Procedure: ArthroFLEX ECM scaffold graft — In patients receiving a graft, thru mini open technique the lateral portal incision will be extended vertically approximately 5-6 cm. A standard, deltoid-splitting, mini-open approach will then be performed, leaving the deltoid attachment to the acromion intact. For arthroscopic technique same method of fixation will be used below. The dermis graft will be sized and cut so as to cover the entire repair site in both medial-lateral and anterior-posterior dimensions.
  Other Names: Surgery with ECM graft
  Arms: Treatment Group
Procedure: Control — This group will undergo rotator cuff repair surgery, but will not receive the ECM scaffold graft.
  Other Names: Surgery without ECM graft
  Arms: Control Treatment Group
Biological: Alternative Treatment Group — Patients who meet pre-op inclusion criteria where a repair cannot be accomplished due to intraoperative findings will remain in the study. This group will be analyzed separately and still follow study procedures.
  Other Names: Repair cannot be accomplished
  Arms: Alternative Treatment Group

SUMMARY:
This trial is to evaluate the effectiveness of the ArthroFLEX® ECM scaffold graph as an augment in rotator cuff repair surgery to reduce the failure rate of rotator cuff repairs for large and massive rotator cuff tears.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled, multi-center clinical trial to evaluate the effectiveness of an ECM scaffold graft to augment repair of a large/massive rotator cuff tear. The study will involve 70 patients. 35 patients will be randomly assigned to each arm of the study.

Despite advances in surgical technology, repairs of large (3-5 cm) and massive (>5 cm) rotator cuff tears (RCT) fail between 20%-90% of the time [1]. Due to their size and increased structural involvement, large or massive RCT present a substantial challenge to orthopaedic surgeons. [16] The repairs tend to fail at the suture-tendon junction, which is due to several factors, including tension at the repair and quality of the tendon [1-2,5]. Full thickness tears are uncommon in younger patients, especially those less than forty years old and are usually traumatic in etiology. Younger patients also typically fair better following arthroscopic rotator cuff repair with fewer failures and more successful return to pre-injury level of function [16]. One strategy to augment repair of large to massive rotator cuff tears has been the development of biological scaffold materials, which are composed of extracellular matrix (ECM). The ECM composing the scaffolds are made from a number of tissues, including, but not limited to, small intestinal submucosa (SIS), dermis, and pericardium [3]. Studies to date include both prospective and retrospective in animal and human models, and include Restore, a porcine-derived SIS by DePuy Orthopaedics, GraftJacket, a human-derived, non-cross-linked dermis graft by Wright Medical Technology, and Zimmer Collagen Repair, a cross-linked porcine derived dermal graft made by Zimmer. Restore studies have shown no benefit and some even an increase in repair failure with recommendations not to use to augment repair. GraftJacket studies have shown a reduction in graft failure; however, several of the Restore and GraftJacket studies are limited by a lack of a control cohort. The Zimmer graft studies have conflicting results with both an improvement and no improvement in failure rates of repair. The prior studies listed are all in vivo; however, the majority are not randomized trials and thus do not have a control with which to compare data. In addition, some trials include open repairs. A lack of prospective, randomized, controlled, in vivo trials exist that evaluate the ability of the ECM scaffold graft augmentation in large to massive arthroscopic rotator cuff repairs to decrease the failure rate.

The purpose of this study is to evaluate the efficacy of using the Arthroflex (A-FLEX) graft to augment large to massive arthroscopic rotator cuff repairs in vivo and decrease repair failures in a prospective, randomized, controlled trial. By undergoing serial US examinations at follow-ups, we also intend to evaluate when during the postoperative period the failure of the repair occurs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a large (2.5-5 cm) to massive (>5 cm) rotator cuff tear who will be undergoing open or arthroscopic repair. The cuff tear size will be determined on either pre-operative magnetic resonance imaging (MRI), or ultrasound (US), or intra-operative measurements, or computerized tomography (CT).
* Patients who are willing and able to provide written informed consent for their involvement in the study.
* Patients who meet criteria for RCR surgery
* Patients older than 18 years of age

Exclusion Criteria:

* Those with a known sensitivity to materials of porcine origin.
* Patients with addiction to illegal drugs, solvents or alcohol who are actively using or have previously attempted and failed a treatment program.
* Patients with bacteremia, a systemic infection, or infection of the surgical site.
* All those who are prisoners.
* Patients who are pregnant or nursing.
* All those with a condition that may limit a patient's ability to finalize the study or that may cause an undue risk to the patient's health and well-being.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory J Gilot, MD, Principal Investigator — Cleveland Clinic Florida
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Derwin KA, Badylak SF, Steinmann SP, Iannotti JP. Extracellular matrix scaffold devices for rotator cuff repair. J Shoulder Elbow Surg. 2010 Apr;19(3):467-76. doi: 10.1016/j.jse.2009.10.020. Epub 2010 Feb 26. PMID 20189415
- [Background] Schlegel TF, Hawkins RJ, Lewis CW, Motta T, Turner AS. The effects of augmentation with Swine small intestine submucosa on tendon healing under tension: histologic and mechanical evaluations in sheep. Am J Sports Med. 2006 Feb;34(2):275-80. doi: 10.1177/0363546505279912. Epub 2005 Oct 6. PMID 16210577
- [Background] Badylak SF, Freytes DO, Gilbert TW. Extracellular matrix as a biological scaffold material: Structure and function. Acta Biomater. 2009 Jan;5(1):1-13. doi: 10.1016/j.actbio.2008.09.013. Epub 2008 Oct 2. PMID 18938117
- [Background] Sclamberg SG, Tibone JE, Itamura JM, Kasraeian S. Six-month magnetic resonance imaging follow-up of large and massive rotator cuff repairs reinforced with porcine small intestinal submucosa. J Shoulder Elbow Surg. 2004 Sep-Oct;13(5):538-41. doi: 10.1016/j.jse.2004.03.005. PMID 15383811
- [Background] Iannotti JP, Codsi MJ, Kwon YW, Derwin K, Ciccone J, Brems JJ. Porcine small intestine submucosa augmentation of surgical repair of chronic two-tendon rotator cuff tears. A randomized, controlled trial. J Bone Joint Surg Am. 2006 Jun;88(6):1238-44. doi: 10.2106/JBJS.E.00524. PMID 16757756
- [Background] Walton JR, Bowman NK, Khatib Y, Linklater J, Murrell GA. Restore orthobiologic implant: not recommended for augmentation of rotator cuff repairs. J Bone Joint Surg Am. 2007 Apr;89(4):786-91. doi: 10.2106/JBJS.F.00315. PMID 17403801
- [Background] Zheng MH, Chen J, Kirilak Y, Willers C, Xu J, Wood D. Porcine small intestine submucosa (SIS) is not an acellular collagenous matrix and contains porcine DNA: possible implications in human implantation. J Biomed Mater Res B Appl Biomater. 2005 Apr;73(1):61-7. doi: 10.1002/jbm.b.30170. PMID 15736287
- [Background] Bond JL, Dopirak RM, Higgins J, Burns J, Snyder SJ. Arthroscopic replacement of massive, irreparable rotator cuff tears using a GraftJacket allograft: technique and preliminary results. Arthroscopy. 2008 Apr;24(4):403-409.e1. doi: 10.1016/j.arthro.2007.07.033. PMID 18375271
- [Background] Badhe SP, Lawrence TM, Smith FD, Lunn PG. An assessment of porcine dermal xenograft as an augmentation graft in the treatment of extensive rotator cuff tears. J Shoulder Elbow Surg. 2008 Jan-Feb;17(1 Suppl):35S-39S. doi: 10.1016/j.jse.2007.08.005. PMID 18201655
- [Background] Soler JA, Gidwani S, Curtis MJ. Early complications from the use of porcine dermal collagen implants (Permacol) as bridging constructs in the repair of massive rotator cuff tears. A report of 4 cases. Acta Orthop Belg. 2007 Aug;73(4):432-6. PMID 17939470
- [Background] Brophy RH, Beauvais RL, Jones EC, Cordasco FA, Marx RG. Measurement of shoulder activity level. Clin Orthop Relat Res. 2005 Oct;439:101-8. doi: 10.1097/01.blo.0000173255.85016.1f. PMID 16205147
- [Background] Parnes N, Bartoszewski NR, Defranco MJ. Arthroscopic Repair of Full-Thickness Rotator Cuff Tears in Active Patients Younger Than 40 Years: 2- to 5-Year Clinical Outcomes. Orthopedics. 2018 Jan 1;41(1):e52-e57. doi: 10.3928/01477447-20171114-02. Epub 2017 Nov 21. PMID 29156071
- [Background] Chung SW, Kim JY, Kim MH, Kim SH, Oh JH. Arthroscopic repair of massive rotator cuff tears: outcome and analysis of factors associated with healing failure or poor postoperative function. Am J Sports Med. 2013 Jul;41(7):1674-83. doi: 10.1177/0363546513485719. Epub 2013 Apr 30. PMID 23631883
- [Background] Greenspoon JA, Petri M, Warth RJ, Millett PJ. Massive rotator cuff tears: pathomechanics, current treatment options, and clinical outcomes. J Shoulder Elbow Surg. 2015 Sep;24(9):1493-505. doi: 10.1016/j.jse.2015.04.005. Epub 2015 Jun 28. PMID 26129871

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Started | 4 | 4 | 1
Completed | 4 | 3 | 1
Not Completed | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group | Total
Number analyzed (Participants) | 4 | 3 | 1 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 0 | 6
  >=65 years | 1 | 0 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.25 (4.57) | 62.66 (2.08) | 76.00 | 63.12 (6.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 1 | 3
  Male | 4 | 1 | 0 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 3
  Not Hispanic or Latino | 2 | 2 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 4 | 2 | 1 | 7
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 1 | 8
American Society of Anesthesiologists (ASA) Physical Status Classification System [Count of Participants; unit: Participants] — The American Society of Anesthesiologists (ASA) 1 category corresponds to a normal healthy patient. A patient categorized as ASA 2 is a patient with mild systemic disease without substantive functional limitations (i.e., well-controlled diabetes or hypertension) while a patient categorized as ASA 3 is a patient with severe systemic disease (i.e., poorly controlled diabetes or hypertension). The higher the ASA number, the worse the physical status of the patient.
  Participants
    ASA 1 | 2 | 0 | 0 | 2
    ASA 2 | 0 | 3 | 1 | 4
    ASA 3 | 2 | 0 | 0 | 2
Smoking Status [Count of Participants; unit: Participants]
  Never Smoked | 4 | 1 | 0 | 5
  Former Smoker | 0 | 2 | 1 | 3
  Smoker | 0 | 0 | 0 | 0
Body Mass Index [Mean (Standard Deviation); unit: Kg/m^2] | 31.36 (2.75) | 31.59 (6.21) | 23.21 | 30.43 (4.77)

OUTCOME MEASURES:

1. Primary Outcome: Tendon Healing
Description: Success as defined by tendon healing after rotator cuff repair, as indicated based on MRI
Time Frame: As assessed 1 year postoperatively.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 3 | 1
Participants | 0 | 3 | 1

2. Primary Outcome: Comparison of Healing by MRI vs US
Description: Comparison of tendon healing will be assessed using US imaging modalities versus MRI (Success as defined by tendon healing after rotator cuff repair, as indicated based on US)
Time Frame: As assessed 1 year postoperatively.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 3 | 1
Participants | 0 | 3 | 1

3. Primary Outcome: Progress of Tendon Healing
Description: Progress of tendon healing based on US will be used as predictive data for 1 year success (based on primary outcome) (Success as defined by tendon healing after rotator cuff repair, as indicated based on US)
Time Frame: As assessed at 6 weeks postoperatively.
Population: Ultrasound was not performed in one patient of the control group
Measure: Count of Participants; unit: Participants
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 3 | 3 | 1
Participants | 3 | 3 | 1

4. Primary Outcome: Progress of Tendon Healing
Description: as for outcome 3
Time Frame: As assessed at 3 months postoperatively.
Population: Ultrasound was not performed in 2 patients of the control group
Measure: Count of Participants; unit: Participants
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 2 | 3 | 1
Participants | 1 | 3 | 1

5. Primary Outcome: Progress of Tendon Healing
Description: as for outcome 3
Time Frame: As assessed at 6 months postoperatively.
Population: Ultrasound was not performed in one patient of the control group
Measure: Count of Participants; unit: Participants
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 3 | 3 | 1
Participants | 3 | 3 | 1

6. Primary Outcome: Progress of Tendon Healing
Description: as for outcome 3
Time Frame: As assessed at 9 months postoperatively.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 3 | 1
Participants | 0 | 3 | 1

7. Secondary Outcome: Patient Outcomes: The American Shoulder and Elbow Surgeon Shoulder Score (ASES)
Description: The ASES is standardized form for assessment of the shoulder. The patient self-evaluation section form contains visual analog scales for pain and activities of daily living questionnaire. The activities of daily living questionnaire is marked on a four-point ordinal scale that can be converted to a cumulative activities of daily living index. A shoulder score can be derived from the visual analogue scale score for pain (50%) and the cumulative activities of daily living score (50%). Scores range from 0 to 100. The higher the score, the better the outcome.
Time Frame: Preoperative
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 3 | 1
Units on a scale | 50.75 (20.15) | 37.66 (15.69) | 52.00

8. Secondary Outcome: Patient Outcomes: The American Shoulder and Elbow Surgeon Shoulder Score (ASES)
Description: as for outcome 7
Time Frame: 6 weeks after surgery
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 3 | 1
Units on a scale | 58.25 (20.20) | 58.66 (21.00) | 45.00

9. Secondary Outcome: Patient Outcomes: The American Shoulder and Elbow Surgeon Shoulder Score (ASES)
Description: as for outcome 7
Time Frame: 3 months after surgery
Population: One patient in the control group and another in the alternative group did not complete the survey
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 3 | 3 | 0
Units on a scale | 66.66 (21.38) | 74.00 (19.05) |

10. Secondary Outcome: Patient Outcomes: The American Shoulder and Elbow Surgeon Shoulder Score (ASES)
Description: as for outcome 7
Time Frame: 6 months after surgery
Population: One patient in the control group and another in the alternative group did not complete the survey
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 3 | 3 | 0
Units on a scale | 73.00 (26.51) | 77.00 (16.52) |

11. Secondary Outcome: Patient Outcomes: The American Shoulder and Elbow Surgeon Shoulder Score (ASES)
Description: as for outcome 7
Time Frame: 9 months after surgery
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 3 | 1
Units on a scale | 82.75 (21.96) | 77.66 (7.50) | 60.00

12. Secondary Outcome: Patient Outcomes: The American Shoulder and Elbow Surgeon Shoulder Score (ASES)
Description: as for outcome 7
Time Frame: 1 year after surgery
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 3 | 1
Units on a scale | 85.00 (15.03) | 88.00 (6.55) | 55.00

13. Secondary Outcome: Patient Outcomes: The Western Ontario Rotator Cuff Index (WORC)
Description: A disease-specific quality of life measurement tool for patients with rotator cuff disease. Patients will respond to by marking a scale with ranges between none and extreme. Information collected includes physical symptoms, such as pain and weakness levels in the shoulder, the impact of the patient's shoulder injury on their sports/recreational activities, work (inside or outside of the home), lifestyle/activities of daily living (ADL), and its emotional impact, such as frustration level, depression, and any worry/concern a patient might be about how their injury might affect their occupation. Total final WORC scores range from 0% to 100%. The higher the score, the better the outcome.
Time Frame: Preoperative
Measure: Mean (Standard Deviation); unit: Percentage of highest functional level
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 3 | 1
Percentage of highest functional level | 34.25 (19.61) | 30.00 (11.26) | 20.00

14. Secondary Outcome: Patient Outcomes: The Western Ontario Rotator Cuff Index (WORC)
Description: as for outcome 13
Time Frame: 6 weeks after surgery
Measure: Mean (Standard Deviation); unit: Percentage of highest functional level
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 3 | 1
Percentage of highest functional level | 63.50 (14.34) | 53.66 (25.92) | 26.00

15. Secondary Outcome: Patient Outcomes: The Western Ontario Rotator Cuff Index (WORC)
Description: as for outcome 13
Time Frame: 3 months after surgery
Population: The patient in the alternative group did not complete the survey
Measure: Mean (Standard Deviation); unit: Percentage of highest functional level
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 3 | 0
Percentage of highest functional level | 64.25 (17.30) | 65.00 (30.64) |

16. Secondary Outcome: Patient Outcomes: The Western Ontario Rotator Cuff Index (WORC)
Description: as for outcome 13
Time Frame: 6 months after surgery
Population: One patient in the control group and another in the alternative group did not complete the survey
Measure: Mean (Standard Deviation); unit: Percentage of highest functional level
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 3 | 2 | 0
Percentage of highest functional level | 65.33 (26.57) | 78.00 (18.38) |

17. Secondary Outcome: Patient Outcomes: The Western Ontario Rotator Cuff Index (WORC)
Description: as for outcome 13
Time Frame: 9 months after surgery
Measure: Mean (Standard Deviation); unit: Percentage of highest functional level
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 3 | 1
Percentage of highest functional level | 71.50 (24.20) | 86.00 (7.00) | 54.00

18. Secondary Outcome: Patient Outcomes: The Western Ontario Rotator Cuff Index (WORC)
Description: as for outcome 13
Time Frame: 1 year after surgery
Measure: Mean (Standard Deviation); unit: Percentage of highest functional level
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 3 | 1
Percentage of highest functional level | 91.50 (15.02) | 94.33 (7.37) | 41.00

19. Secondary Outcome: Patient Outcomes: Measurement of Shoulder Activity Level
Description: This activity scale was developed using established principles: item generation, item reduction, pretesting, and reliability and validity testing. The activity rating is a numerical sum of scores for five activities rated on a five-point frequency scale from never performed (0 points) to daily (4 points). Patients were scored on the following criteria: carrying an object 8 lb or heavier by hand, handling objects overhead, weight training with arms, swinging motion (i.e., hitting tennis or golf ball), and lifting objects 25 lb or heavier. It can be used in conjunction with patient-based measures of shoulder outcome to define patient populations for cohort studies, and to assess activity level as a prognostic factor in patients with shoulder disorders. Scores range from 0 to 20. The higher the score, the better the outcome.
Time Frame: Preoperative
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 3 | 1
Units on a scale | 4.75 (5.25) | 2.00 (2.64) | 3.00

20. Secondary Outcome: Patient Outcomes: Measurement of Shoulder Activity Level
Description: as for outcome 19
Time Frame: 6 weeks after surgery
Population: One patient in the treatment group did not complete the survey
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 2 | 1
Units on a scale | 2.25 (1.70) | 8.50 (12.02) | 14.00

21. Secondary Outcome: Patient Outcomes: Measurement of Shoulder Activity Level
Description: as for outcome 19
Time Frame: 3 months after surgery
Population: The patient in the alternative group did not complete the survey
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 3 | 0
Units on a scale | 8.25 (6.65) | 4.66 (7.23) |

22. Secondary Outcome: Patient Outcomes: Measurement of Shoulder Activity Level
Description: as for outcome 19
Time Frame: 6 months after surgery
Population: One patient in the control group did not complete the survey
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 3 | 3 | 1
Units on a scale | 10.66 (8.14) | 10.66 (9.01) | 9.00

23. Secondary Outcome: Patient Outcomes: Measurement of Shoulder Activity Level
Description: as for outcome 19
Time Frame: 9 months after surgery
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 3 | 1
Units on a scale | 7.50 (6.55) | 12.00 (4.00) | 2.00

24. Secondary Outcome: Patient Outcomes: Measurement of Shoulder Activity Level
Description: as for outcome 19
Time Frame: 1 year after surgery
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 3 | 1
Units on a scale | 12.50 (5.80) | 11.33 (8.50) | 0.00

25. Secondary Outcome: Patient Outcomes: Subjective Shoulder Value (SSV)
Description: The SSV is defined as a patient's subjective shoulder assessment expressed as a percentage of an entirely normal shoulder, which would score 100%. Scores range from 0 to 100. The higher the score, the better the outcome.
Time Frame: Preoperative
Measure: Mean (Standard Deviation); unit: percentage of entirely normal shoulder
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 3 | 1
percentage of entirely normal shoulder | 32.50 (5.00) | 36.66 (15.27) | 20.00

26. Secondary Outcome: Patient Outcomes: Subjective Shoulder Value (SSV)
Description: as for outcome 25
Time Frame: 6 weeks after surgery
Measure: Mean (Standard Deviation); unit: percentage of entirely normal shoulder
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 3 | 1
percentage of entirely normal shoulder | 57.75 (40.08) | 60.00 (20.00) | 40.00

27. Secondary Outcome: Patient Outcomes: Subjective Shoulder Value (SSV)
Description: as for outcome 25
Time Frame: 3 months after surgery
Population: The patient in the alternative group did not complete the survey
Measure: Mean (Standard Deviation); unit: percentage of entirely normal shoulder
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 3 | 0
percentage of entirely normal shoulder | 76.25 (12.50) | 78.33 (12.58) |

28. Secondary Outcome: Patient Outcomes: Subjective Shoulder Value (SSV)
Description: as for outcome 25
Time Frame: 6 months after surgery
Population: One patient in the control group and another in the treatment group did not complete the survey
Measure: Mean (Standard Deviation); unit: percentage of entirely normal shoulder
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 3 | 2 | 1
percentage of entirely normal shoulder | 71.66 (22.54) | 82.50 (10.60) | 75.00

29. Secondary Outcome: Patient Outcomes: Subjective Shoulder Value (SSV)
Description: as for outcome 25
Time Frame: 9 months after surgery
Measure: Mean (Standard Deviation); unit: percentage of entirely normal shoulder
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 3 | 1
percentage of entirely normal shoulder | 72.50 (26.29) | 83.33 (15.27) | 80.00

30. Secondary Outcome: Patient Outcomes: Subjective Shoulder Value (SSV)
Description: as for outcome 25
Time Frame: 1 year after surgery
Measure: Mean (Standard Deviation); unit: percentage of entirely normal shoulder
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 3 | 1
percentage of entirely normal shoulder | 85.75 (14.56) | 91.66 (2.88) | 75.00

31. Secondary Outcome: Patient Outcomes: Constant Score (CS)
Description: C Constant and A Murley. This scoring system consists of four variables that are used to assess the function of the shoulder. The right and left shoulders are assessed separately. The subjective variables are pain and ADL (sleep, work, recreation / sport) which give a total of 35 points. Constant subjective scale goes from 0 to 35. The higher the score, the better the outcome.
Time Frame: Preoperative
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 3 | 1
Units on a scale | 12.75 (3.59) | 10.66 (6.65) | 9.00

32. Secondary Outcome: Patient Outcomes: Constant Score (CS)
Description: as for outcome 31
Time Frame: 6 weeks after surgery
Population: One patient in the control group did not complete the survey
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 3 | 3 | 1
Units on a scale | 18.33 (0.57) | 15.00 (2.64) | 13.00

33. Secondary Outcome: Patient Outcomes: Constant Score (CS)
Description: as for outcome 31
Time Frame: 3 months after surgery
Population: The patient in the alternative group did not complete the survey
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 3 | 0
Units on a scale | 20.00 (3.55) | 18.00 (3.46) |

34. Secondary Outcome: Patient Outcomes: Constant Score (CS)
Description: as for outcome 31
Time Frame: 6 months after surgery
Population: One patient in the control group did not complete the survey
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 3 | 3 | 1
Units on a scale | 18.00 (5.56) | 21.33 (4.16) | 27.00

35. Secondary Outcome: Patient Outcomes: Constant Score (CS)
Description: as for outcome 31
Time Frame: 9 months after surgery
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 3 | 1
Units on a scale | 21.00 (6.97) | 20.33 (0.57) | 14.00

36. Secondary Outcome: Patient Outcomes: Constant Score (CS)
Description: as for outcome 31
Time Frame: 1 year after surgery
Population: One patient in the control group did not complete the survey
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 3 | 3 | 1
Units on a scale | 20.33 (4.50) | 15.66 (4.50) | 15.00

37. Secondary Outcome: The Veterans RAND 12 Item Health Survey (VR-12) (Physical Component Score)
Description: The Veterans RAND 12 Item Health Survey (VR-12) was designed to replicate much of the behavior of the Veterans RAND 36 Item Health Survey (VR-36) with a reduced number of questions. The results of the VR-12 are summarized as two scores - a Mental Component Score (MCS) and a Physical Component Score (PCS). These summary scores range from 0 to 100. The higher the score, the better the outcome.
Time Frame: Preoperative
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 3 | 1
Units on a scale | 42.50 (3.10) | 39.33 (6.50) | 38.00

38. Secondary Outcome: The Veterans RAND 12 Item Health Survey (VR-12) (Physical Component Score)
Description: as for outcome 37
Time Frame: 6 weeks after surgery
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 3 | 1
Units on a scale | 43.00 (6.68) | 43.33 (4.16) | 37.00

39. Secondary Outcome: The Veterans RAND 12 Item Health Survey (VR-12) (Physical Component Score)
Description: as for outcome 37
Time Frame: 3 months after surgery
Population: One patient in the treatment group and another in the alternative group did not complete the survey
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 2 | 0
Units on a scale | 52.50 (1.29) | 45.50 (12.02) |

40. Secondary Outcome: The Veterans RAND 12 Item Health Survey (VR-12) (Physical Component Score)
Description: as for outcome 37
Time Frame: 6 months after surgery
Population: One patient in the control group did not complete the survey
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 3 | 3 | 1
Units on a scale | 48.66 (9.60) | 50.00 (8.71) | 49.00

41. Secondary Outcome: The Veterans RAND 12 Item Health Survey (VR-12) (Physical Component Score)
Description: as for outcome 37
Time Frame: 9 months after surgery
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 3 | 1
Units on a scale | 53.00 (8.71) | 50.66 (3.78) | 48.00

42. Secondary Outcome: The Veterans RAND 12 Item Health Survey (VR-12) (Physical Component Score)
Description: as for outcome 37
Time Frame: 1 year after surgery
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 3 | 1
Units on a scale | 57.25 (3.50) | 54.33 (8.38) | 37.00

43. Secondary Outcome: The Veterans RAND 12 Item Health Survey (VR-12) (Mental Component Score)
Description: as for outcome 37
Time Frame: Preoperative
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 3 | 1
Units on a scale | 43.50 (8.34) | 37.66 (19.85) | 53.00

44. Secondary Outcome: The Veterans RAND 12 Item Health Survey (VR-12) (Mental Component Score)
Description: as for outcome 37
Time Frame: 6 weeks after surgery
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 3 | 1
Units on a scale | 48.00 (7.34) | 31.33 (4.50) | 59.00

45. Secondary Outcome: The Veterans RAND 12 Item Health Survey (VR-12) (Mental Component Score)
Description: as for outcome 37
Time Frame: 3 months after surgery
Population: One patient in the treatment group and another in the alternative group did not complete the survey
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 2 | 0
Units on a scale | 37.75 (5.67) | 38.50 (2.12) |

46. Secondary Outcome: The Veterans RAND 12 Item Health Survey (VR-12) (Mental Component Score)
Description: as for outcome 37
Time Frame: 6 months after surgery
Population: One patient in the control group did not complete the survey
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 3 | 3 | 1
Units on a scale | 47.00 (9.84) | 33.66 (11.84) | 41.00

47. Secondary Outcome: The Veterans RAND 12 Item Health Survey (VR-12) (Mental Component Score)
Description: as for outcome 37
Time Frame: 9 months after surgery
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 3 | 1
Units on a scale | 40.25 (9.50) | 33.33 (5.85) | 47.00

48. Secondary Outcome: The Veterans RAND 12 Item Health Survey (VR-12) (Mental Component Score)
Description: as for outcome 37
Time Frame: 1 year after surgery
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
Number analyzed (Participants) | 4 | 3 | 1
Units on a scale | 37.25 (9.77) | 33.66 (9.07) | 53.00

ADVERSE EVENTS:
Time Frame: Within 1 year after surgery
Arm/Group | Control Treatment Group | Treatment Group | Alternative Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 3/4 | 1/3 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Treatment Group (N=4) | Treatment Group (N=3) | Alternative Treatment Group (N=1)
Dry eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Posterior vitrous detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Pain from shoulder to hand (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Low back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Atypical chest pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Back muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Foot pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hip contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Shoulder tear (contralateral) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Covid-19 positive (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/09/NCT03551509/Prot_SAP_000.pdf